CLINICAL TRIAL: NCT00735085
Title: A Randomized, Double Blind, Placebo-Controlled Dose Escalation Study to Investigate the Safety and Pharmacokinetics After Single and Multiple Doses of SLV334 in Sequential Cohorts of Patients With Moderate and Severe Traumatic Brain Injury
Brief Title: A Phase 2a Dose Escalation Study With SLV334 in Patients With Traumatic Brain Injury.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was stopped 20 May 2010 due to strategic considerations
Sponsor: Abbott Products (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S334.2.002; 2008-001409-40 (EudraCT Number)
Record Dates: First submitted 2007-11-30; First posted 2008-08-14 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SLV334 (Experimental)
  Interventions: Drug: SLV334
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLV334 — 1000mg SLV334 as a single dose
  Arms: SLV334
Drug: SLV334 — 1000mg SLV334 b.i.d. for one day
  Arms: SLV334
Drug: SLV334 — 2000mg SLV334 b.i.d. for one day
  Arms: SLV334
Drug: SLV334 — 2000mg SLV334 b.i.d. for three days
  Arms: SLV334
Drug: Placebo — SLV334 Placebo arm
  Arms: Placebo

SUMMARY:
A Randomized, Double Blind, Placebo Controlled, Phase 2 Dose Escalation Study to Investigate the Safety and Pharmacokinetics after Single and Multiple I.V. Doses of SLV334 in Sequential Cohorts of Patients with Moderate and Severe Traumatic Brain Injury.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients, age between 16 and 70 years, inclusive.
2. Sustained a closed [non-penetrating] head trauma no more than 8 hours before initiation of drug treatment with study drug at the study hospital;
3. TBI diagnosed by history, clinical examination with GCS of 12 or less.
4. Evidence of TBI confirmed by abnormalities on CT scan
5. Clinical indication to monitor ICP
6. Informed consent is given.

Exclusion Criteria

1. Any spinal cord injury;
2. Pregnant or lactating women;
3. Patients with penetrating head injury;
4. Bilaterally fixed dilated pupils at the time of randomization;
5. Coma suspected to be primarily due to other causes than head injury such as drug or alcohol overdose;
6. Severe multiple trauma or major organ failure (uncontrolled visceral bleeding, unstable cardio-respiratory or renal function);
7. Known treatment with another investigational drug therapy within 30 days of injury.
8. Life expectancy of less than 24 hours.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety of SLV334 including mortality, adverse events (AE), serious adverse events (SAE), vitals signs, laboratory variables and ECG | 2 weeks

SECONDARY OUTCOMES:
PK parameters of SLV334 | up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Bronzowa, MD, Study Director — Abbott Products
Locations (14):
- United States (5):
  - Site Reference ID/Investigator# 45771, Baltimore, Maryland
  - Site Reference ID/Investigator# 45775, Dayton, Ohio
  - Site Reference ID/Investigator# 45770, Portland, Oregon
  - Site Reference ID/Investigator# 45785, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 45780, Pittsburgh, Pennsylvania
- Israel (4):
  - Site Reference ID/Investigator# 45727, Haifa
  - Site Reference ID/Investigator# 45726, Jerusalem
  - Site Reference ID/Investigator# 45723, Ramat Gan
  - Site Reference ID/Investigator# 45725, Tel Aviv
- Italy (2):
  - Site Reference ID/Investigator# 45735, Milan
  - Site Reference ID/Investigator# 45731, Monza
- Spain (3):
  - Site Reference ID/Investigator# 45765, Barcelona
  - Site Reference ID/Investigator# 45762, Madrid
  - Site Reference ID/Investigator# 45763, Palma de Mallorca